CLINICAL TRIAL: NCT05391529
Title: Patients Decision Making in Choosing Between Colonic Investigation Alternatives
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Highland (Other)
Responsible Party: Sponsor
Other Study IDs: 2-014-22
Record Dates: First submitted 2022-04-11; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colonoscopy: Patients awaiting colonoscopy
  Interventions: Behavioral: Interview
- CCE: Patients awaiting colon capsule endoscopy
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Semi structured patient interview via telephone

SUMMARY:
This is a qualitative interview study to understand patients' priorities for different aspects of tests when considering a colonic investigation. Patients currently waiting for colon capsule endoscopy (CCE), and colonoscopy will be invited to take part. Semi-structured interviews will be carried out over the telephone following an interview guide. Recorded interviews will be transcribed and undergo thematic analysis. We will seek to publish the results of this study to inform future research and developments for colonic investigations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 who are on the waiting list for a colonoscopy or CCE. Only patients who can provide valid consent will be included.
* English language speaking (translation services are not available for this study).

Exclusion Criteria:

* Patients undergoing colonoscopy due to positive bowel screening test or due to surveillance of known colonic pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve recruiting patients on the waiting list for colonoscopy or colon capsule endoscopy from one NHS Scotland Health Board.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Completion of a qualitative interview discussing the patients priorities for different aspects of tests when considering a colonic investigation | Through study completion, an average of 6 months
  We will invite patients to undergo qualitative telephone interviews to establish their priorities for different aspects of tests when considering a colonic investigation.

SECONDARY OUTCOMES:
Completion of a qualitative interview discussing what patients' perceptions of the decision-making process are when choosing between colonic investigations | Through study completion, an average of 6 months
  We will invite patients to undergo qualitative telephone interviews to establish their perceptions of the decision making process when choosing between colonic investigations.

IPD SHARING:
Plan to Share IPD: No
This is a qualitative interview study so individual data will not be available to share

REFERENCES:
- [Derived] MacLeod C, Treweek S, Wilson P, Watson AJM, Robinson S. Patient priorities and decision-making process when choosing between colonic investigation alternatives: a qualitative interview study. BMJ Open Gastroenterol. 2025 Aug 22;12(1):e001602. doi: 10.1136/bmjgast-2024-001602. PMID 40846494